CLINICAL TRIAL: NCT00205959
Title: Comparison of Standard Treatment Methods for Proximal Humerus Fractures
Brief Title: LPHP-Philos-PHN Conservative Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry); AO Research Fund (Other)
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-LPP-04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Proximal Humeral Fracture
Keywords: Humerus; Fractures; Locking Plates; Nail System
MeSH Terms: conditions — Shoulder Fractures; Fractures, Bone

INTERVENTIONS:
Device: Locking proximal humerus plate
Device: Proximal Humerus Internal Locking System
Device: Proximal Humerus Nail

SUMMARY:
The aim of the study is to compare the results regarding fracture healing

and functional outcome after the treatment of proximal humeral fractures

with the four different treatment methods after 12w./6months and 12 months

based on radiological evaluation as well as the "constant score" and the

"neer score".

DETAILED DESCRIPTION:
Evaluation of proximal humeral fractures using a new stable-angled implant.

ELIGIBILITY:
Inclusion Criteria:

* fractures of proximal humerus
* age over 18 years
* completed skeletal development
* fracture less than 5 days old

Exclusion Criteria:

* open fractures
* pseudoarthrosis, pathological or refractures
* ipsilateral fractures of distal humerus or elbow
* polytraumatic conditions
* pregnancy
* subject with known history of diseases that influence the healing process
* alcohol, drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640
Dates: Start 2002-08; Study Completion 2006-08

PRIMARY OUTCOMES:
Radiological comparison of the fracture healing
Functional outcome based on "constant and neer score" after 12 months

SECONDARY OUTCOMES:
Analysis of occured complications
Radiological evaluation of possible misallocation
Subjective patient judgement of before and after treatment according to DASH-questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Südkamp, Prof. MD, Principal Investigator — Universitaetsklinik Freiburg
Locations (1):
- Universitaestklinik Freiburg, Klinik für Traumatologie, Freiburg im Breisgau, Germany